CLINICAL TRIAL: NCT00686855
Title: An Open Label Phase II Randomized Trial of Topical Dexamethasone and Tacrolimus for the Treatment of Oral Chronic Graft-Versus-Host Disease
Brief Title: Topical Dexamethasone and Tacrolimus for the Treatment of Oral Chronic Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Boston Children's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Nathaniel S. Treister, DMD, DMSc, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-027
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2014-02-19 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: Oral Chronic Graft-versus-host Disease
Keywords: tacrolimus; dexamethasone; oral rinse
MeSH Terms: interventions — Tacrolimus; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Experimental): Tacrolimus Arm Closed to Accrual as of January 2012
  Interventions: Drug: Tacrolimus
- Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus elixir taken as an oral rinse four times a day for 4 weeks
  Arms: Tacrolimus
Drug: Dexamethasone — Dexamethasone elixir taken as an oral rinse 4 times a day for 4 weeks
  Arms: Dexamethasone

SUMMARY:
The purpose of this research study is to determine the effectiveness of topical steroid therapy (with a drug called dexamethasone) and topical tacrolimus therapy for the treatment of oral chronic Graft-Versus-Host Disease (cGVHD)

DETAILED DESCRIPTION:
* Because no one knows which study option is best, participants will be "randomized" into one of two study groups: topical dexamethasone or topical tacrolimus.
* Participants will take the medication by mouth rinse four times a day for 5 minutes at a time. After rinsing they will spit out the medication and will not be able to eat or drink for 15 minutes.
* Participants will also take anti-fungal medication (fluconazole) orally once a week.
* After two weeks on study treatment, participants will have a blood drawn to monitor tacrolimus levels.
* After the final treatment (4 weeks), participants will have the following tests and procedures: clinical examination; questionnaire; blood tests; oral culture; optional tissue biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oral chronic graft-versus-host disease
* Patients 4 years of age or older
* Stable cGVHD medication regimen for the four weeks prior to study enrollment

Exclusion Criteria:

* Patients already on topical steroid or tacrolimus therapies

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-08; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Treister, DMD, Principal Investigator — Brigham and Women's Hospital
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone: Dexamethasone : Dexamethasone elixir taken as an oral rinse 4 times a day for 4 weeks
- Tacrolimus: Tacrolimus Arm Closed to Accrual as of January 2012
  Tacrolimus : Tacrolimus elixir taken as an oral rinse four times a day for 4 weeks
Period: Overall Study
Arm/Group | Dexamethasone | Tacrolimus
Started | 28 | 18
Completed | 27 | 17
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Progressive GVHD | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Tacrolimus | Total
Number analyzed (Participants) | 28 | 18 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 12 | 34
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (11.5) | 54.9 (15.3) | 54.2 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 6 | 23
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 28 | 18 | 46

OUTCOME MEASURES:

1. Primary Outcome: The Clinical Efficacy of Topical Steroid and Topical Tacrolimus Therapies for the Treatment of Oral cGHVD.
Description: Participants were given a survey at the time of screening and 4 weeks after start of therapy. The participants self-reported three symptoms of oral cGVHD: oral sensitivity, mouth pain, and mouth dryness. Each symptom was given a score ranging from 0-10, with 0 as none and 10 as the worst. Improvement in subjective scores was defined as 3 points or further reduction from pre-treatment to post-treatment assessment.
Time Frame: Participants were assessed at Baseline and 4 weeks after start of therapy
Population: Of the 46 participants enrolled on the trial, 36 were deemed evaluable for response.
Measure: Number; unit: participants
Arm/Group | Dexamethasone | Tacrolimus
Number analyzed (Participants) | 22 | 14
participants
  Improvement in Oral Sensitivity | 15 | 3
  Improvement in Mouth Pain | 11 | 2
  Improvement in Mouth Dryness | 11 | 5
  Improvement in 1 or more areas | 17 | 7
  Improvement in 2 or more areas | 13 | 2
  Improvement in all 3 areas | 7 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the four week peroid participants took the study treatment.
Arm/Group | Dexamethasone | Tacrolimus
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/18
Other Adverse Events (participants affected / at risk) | 1/28 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=28) | Tacrolimus (N=18)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — deemed unrelated to study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 3.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=28) | Tacrolimus (N=18)
Pain - Oral Cavity (General disorders) | 1 (1) | 0 (0)
Infection Gr0-2 neutrophils - oral cavity (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes